CLINICAL TRIAL: NCT04955795
Title: Telemedicine for Unhealthy Alcohol Use in Persons Living With HIV Using Common Elements Treatment Approach
Brief Title: Telemedicine for Unhealthy Alcohol Use in Persons Living With HIV Using CETA
Acronym: TALC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Karen Cropsey, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300007410; P01AA029540 (NIH)
Record Dates: First submitted 2021-05-26; First posted 2021-07-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Hiv; Alcohol Problem
Keywords: HIV Outcomes; Unhealthy Alcohol Use; Mental Health; Medication Adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol-Related Disorders; Psychological Well-Being; Medication Adherence | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol Brief Intervention (BI) (Active Comparator): At the time of trial enrollment, participants will receive a session of alcohol brief intervention (BI) via telephone.
  Interventions: Behavioral: Alcohol Brief Intervention (BI)
- Common Elements Treatment Approach (CETA) via Telemedicine (Experimental): Participants will be provided with 6 to 12 weekly CETA sessions via telephone.
  Interventions: Behavioral: Alcohol Brief Intervention (BI); Behavioral: Common Elements Treatment Approach (CETA) via Telemedicine

INTERVENTIONS:
Behavioral: Alcohol Brief Intervention (BI) — The BI we will use was based on CETA's substance use module and was designed for one-on-one delivery. It is comprised of 6 elements (i.e. assessment, understanding impacts, exploring change, goal setting, identifying the reasons, and skill building) including a 2-week alcohol timeline follow back assessment, which is completed by the therapist. BI will be provided by a trained research assistant who has completed consent, enrollment, and randomized procedures with the client.
Behavioral: Common Elements Treatment Approach (CETA) via Telemedicine — CETA consists of nine key elements (i.e. engagement and education; safety assessment and planning; psychoeducation/introduction; substance use reduction; behavioral activation; cognitive coping/restructuring; relaxation; exposure; and problem solving) that address common mental health problems such as trauma, PTSD, depression, and anxiety. Participants randomized to CETA will be assigned to a CETA provider (clinical psychology or social work graduate student or master's degree substance abuse counselor). Enrolled participants will be discussed at weekly supervision meetings. An individualized treatment plan will be designed for each participant including type and order of CETA modules. The counselor will contact the participant by phone to schedule CETA sessions and follow up any missed appointments. Counselors, who will also be given a unique ID# for documentation and analysis, will carry 3-10 active CETA cases at a time depending on their experience level.
  Arms: Common Elements Treatment Approach (CETA) via Telemedicine

SUMMARY:
This study is designed to examine the efficacy of a brief intervention plus a cognitive-behavioral intervention compared to brief intervention alone to address unhealthy alcohol use and comorbid mental health symptoms to improve HIV outcomes among people living with HIV in Alabama.

DETAILED DESCRIPTION:
Participants will be randomly assigned to receive either Alcohol Brief Intervention (BI) or BI plus Common Elements Treatment Approach (T-CETA) via telephone. Participants will receive either 1 phone session of BI or 6 to 12 weekly phone sessions of BI + T-CETA. Follow ups will occur at 6 and 12 months with participants.

Participants will provide data on alcohol use, mental health comorbidities, HIV outcomes, medication adherence, and laboratory collections (CD4+ T cell count, viral load, and an alcohol biomarker: PEth) at the baseline assessment and again at the 6 and 12 month follow ups.

The study will also conduct mixed methods implementation measures with a subset of participants who are selected across various strata (i.e. gender, age, trial arm).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Living with HIV infection
* Receiving HIV care at 1 of 4 participating AQMG sites (Alabama Quality Management Group sites - i.e. Ryan White HIV/AIDS Program-funded community clinics in Alabama)
* Unhealthy alcohol use documented on the AUDIT survey delivered via PRO (i.e. 4 or greater points for women and greater than 8 points for men).

Exclusion Criteria:

* Inability to use a mobile phone due to cognitive or physical impairments
* Unable to speak sufficient English to provide informed consent and receive cognitive behavioral therapy
* Active suicidality or psychosis
* Risk for acute alcohol withdrawal or seizures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Alcohol Use at 6 months | 6 months
  Defined by the participant's score on the Alcohol Use Disorders Identification Test (AUDIT). The minimum score on the AUDIT measure is 0, and the maximum score on the AUDIT measure is 40. For women, a score of of 4 or greater indicates hazardous or harmful alcohol consumption. For men, a score of 8 or greater indicates hazardous or harmful alcohol consumption. Higher scores on the AUDIT measure indicates more hazardous or harmful alcohol consumption.
Change from Baseline Alcohol Use at 6 months | 6 months
  Defined by the participant's blood level of phosphatidylethanol (PEth). Participants will undergo a finger prick to collect a blood sample which will be analyzed for PEth level. PEth level of less than 20 ng/mL indicates abstinence or light drinking (from not drinking to averaging less than two drinks/day for several days a week). PEth level of 20-200 ng/mL indicates moderate level of drinking (averaging between 2 to 4 drinks/day for several days a week). Higher levels of PEth in the blood indicate more hazardous or harmful alcohol consumption.

SECONDARY OUTCOMES:
Change from Baseline Substance Use at 6 months | 6 months
  Defined by the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST). The minimum score on each substance (i.e. tobacco, alcohol, cannabis, cocaine, amphetamines, inhalants, sedatives, hallucinogens, opioids, or other substances) is 0 to 3 (Low health risk). Moderate health risk is defined as a score of 4-26. High heath risk is defined as a score of 27 and higher. Higher scores indicate greater risk for health issues as a result of substance use.
Change from Baseline Substance Use at 12 months | 12 months
  Defined by the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST). The minimum score on each substance (i.e. tobacco, alcohol, cannabis, cocaine, amphetamines, inhalants, sedatives, hallucinogens, opioids, or other substances) is 0 to 3 (Low health risk). Moderate health risk is defined as a score of 4-26. High heath risk is defined as a score of 27 and higher. Higher scores indicate greater risk for health issues as a result of substance use.
Change from Baseline Depression at 6 months | 6 months
  Defined by the Patient Health Questionnaire-9 (PHQ9) validated tool. The minimum score on this measure is 0 and the maximum score on this measure is 27. Higher scores on this measure indicates a worse outcome.
Change from Baseline Depression at 12 months | 12 months
  Defined by the Patient Health Questionnaire-9 (PHQ9) validated tool. The minimum score on this measure is 0 and the maximum score on this measure is 27. Higher scores on this measure indicate a worse outcome.
Change from Baseline Anxiety at 6 months | 6 months
  Defined by the Generalized Anxiety Disorder-7 Item (GAD-7) validated tool. The minimum score of this measure is 0, and the maximum score of this measure is 21. Higher scores on this measure indicate a worse outcome.
Change from Baseline Anxiety at 12 months | 12 months
  Defined by the Generalized Anxiety Disorder-7 Item (GAD-7) validated tool. The minimum score of this measure is 0, and the maximum score of this measure is 21. Higher scores on this measure indicate a worse outcome.
Change from Baseline Traumatic Stress at 6 months | 6 months
  Defined by the Post-Traumatic Stress Disorder (PTSD) Checklist for DSM-IV (PCL-4) validated tool. The minimum score of this measure is 0, and the maximum score of this measure is 80. Higher scores on this measure indicate a worse outcome.
Change from Baseline Traumatic Stress at 12 months | 12 months
  Defined by the Post-Traumatic Stress Disorder (PTSD) Checklist for DSM-IV (PCL-4) validated tool. The minimum score of this measure is 0, and the maximum score of this measure is 80. Higher scores on this measure indicate a worse outcome.
Change from Baseline HIV Suppression at 6 months | 6 months
  Defined by Viral Load <20 copies per mL. This testing will be done by the participant's physician and reported to study staff.
Change from Baseline HIV Suppression at 12 months | 12 months
  Defined by Viral Load <20 copies per mL. This testing will be done by the participant's physician and reported to study staff.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cropsey, Psy.D., Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - Health Service Center, Anniston, Alabama
  - UAB Family Clinic, Birmingham, Alabama
  - Thrive, Huntsville, Alabama
  - Five Horizons, Montgomery, Alabama
  - Unity Wellness, Opelika, Alabama

IPD SHARING:
Plan to Share IPD: No